CLINICAL TRIAL: NCT07213934
Title: WOPPPR: Window of Opportunity Phase I and Phase II Trial Combining PD-1 Inhibition and Neoadjuvant Proton or Photon Radiation Therapy in Recurrent Head and Neck Squamous Cell Carcinoma
Brief Title: Phase I/ II Trial Combining PD-1 Inhibition and Neoadjuvant Proton or Photon Radiation Therapy in Recurrent Head and Neck Squamous Cell Carcinoma
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Cincinnati (Other)
Responsible Party: Principal Investigator, Trisha Wise-Draper, Principal Investigator, University of Cincinnati
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UCCC-HN-24-01
Record Dates: First submitted 2025-09-30; First posted 2025-10-09 (Actual); Last update posted 2025-10-15 (Actual); Status verified 2025-10

CONDITIONS: Head and Neck Cancer; Recurrent Head and Neck Squamous Cell Carcinoma
MeSH Terms: conditions — Head and Neck Neoplasms; Squamous Cell Carcinoma of Head and Neck | interventions — Proton Therapy; pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Standard Radiation Therapy (Active Comparator): XRT followed by PD-1 inhibition
  Interventions: Drug: Pembrolizumab
- Photon Therapy (Experimental): PT followed by PD-1 inhibition
  Interventions: Radiation: Proton therapy; Drug: Pembrolizumab

INTERVENTIONS:
Radiation: Proton therapy — Proton therapy is a type of radiation therapy that uses protons rather than x-rays. It painlessly delivers radiation to treat some types of cancer.
  Arms: Photon Therapy
Drug: Pembrolizumab — PDL-1 immunotherapy drug

SUMMARY:
The purpose of the Phase I study is to see if it is safe to use X-ray photon radiation (XRT) and proton radiation (PT) before surgery in patients with recurrent head and neck squamous cell carcinoma (rHNSCC).

The purpose of the Phase II study is to see if using XRT or PT before immunotherapy (pembrolizumab) prior to surgery benefits patients with recurrent head and neck squamous cell carcinoma (rHNSCC).

DETAILED DESCRIPTION:
In phase I, cohorts of 3 to 6 patients will be treated with 3 fractions of RT prior to surgery. A de-escalation cohort is planned if toxicity is exceeded in Cohort 1. The types of RT (XRT and PT) will be tested sequentially. The first cohort will include XRT followed by salvage surgery and adjuvant immunotherapy. The RP2D or dose found to be safe will be decided for XRT first. The RP2D for XRT will then be the starting dose cohort for PT to ensure the dose remains safe. The highest dose found to be safe for both types of RT will be used for Phase II. The dose escalation criteria must be met at each dose level including up to 28 days post-surgical resection in order to enroll and treat pts for phase II or de-escalate to the indicated dose level.

Phase II is a two arm window of opportunity multi-center study investigating XRT or PT with PD-1 inhibition in recurrent HNSCC. The study will be conducted in two stages with 2 independent experimental arms based on a Simons 2 Stage Design. PT followed by PD-1 inhibition (Arm 1) or XRT followed by PD-1 inhibition (Arm 2) will be independently compared to a historical control group with the primary endpoint of major pathological response (MPR) and a goal of 35% of patients achieving MPR compared to a baseline of 10% with PD-1 alone. Forty total patients with recurrent HNSCC will be screened and randomized to avoid selection bias to either PT or XRT. Based on a Simon Stage 2 Design, nine patients are required for stage I. Stage II will proceed after determination of Stage I MPR.

ELIGIBILITY:
Inclusion Criteria (Both Phase I and Phase II)

1. Patients must have histologically or cytologically confirmed recurrent head and neck squamous cell carcinoma including oral cavity, laryngeal, hypopharyngeal, or oropharyngeal (HPV-) SCC.
2. Patients must be a candidate for salvage surgical resection.
3. Patients must have failed prior RT >6 months prior to recurrence with at least 30 Gy delivered to the current target volume.
4. Disease must be limited to a single site or adjacent sites that can be treated in a single contiguous target volume for which the maximum total tumor dimension (GTV) must be <7 cm.
5. Patients must have a CPS PD-L1 of ≥1%. This may be tested on a new biopsy or archival tissue.
6. Age ≥18 years.
7. ECOG performance status ≤1 (or Karnofsky ≥70%, see Appendix A).
8. Patients must have adequate organ and marrow function as defined below:

   Platelets ≥100,000/mcL Total bilirubin ≤ institutional upper limit of normal (ULN) AST(SGOT)/ALT(SGPT) ≤3 × institutional ULN Creatinine ≤ 1.5x institutional upper limit of normal (ULN) OR glomerular filtration rate (GFR) ≥30 mL/min/1.73 m2 (see Appendix B).
9. Archival tissue must be available for baseline analysis. Either a tumor block or at least 20 slides must be available.
10. Known human immunodeficiency virus (HIV)-infected patients on effective anti-retroviral therapy with undetectable viral load within 6 months are eligible for this trial.
11. For patients with evidence of chronic hepatitis B virus (HBV) infection, the HBV viral load must be undetectable on suppressive therapy, if indicated.
12. Patients with a history of hepatitis C virus (HCV) infection must have been treated and cured. For patients with known HCV infection who are currently on treatment, they are eligible if they have an undetectable HCV viral load.
13. Patients with a prior or concurrent malignancy whose natural history or treatment does not have the potential to interfere with the safety or efficacy assessment of the investigational regimen are eligible for this trial.
14. Patients with known history or current symptoms of cardiac disease, or history of treatment with cardiotoxic agents, should have a clinical risk assessment of cardiac function using the New York Heart Association Functional Classification. To be eligible for this trial, patients should be class 2B or better.
15. Women of child-bearing potential and men must agree to use adequate contraception (e.g., hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately. Men treated or enrolled on this protocol must also agree to use adequate contraception prior to the study, for the duration of study participation, and for 4 months after completion of pembrolizumab administration.
16. Ability to understand and the willingness to sign a written informed consent document. Legally authorized representatives may sign and give informed consent on behalf of study participants.

Exclusion Criteria (Phase I & II)

1. Patients who have metastatic disease.
2. Patients who have ongoing adverse events from prior anti-cancer therapy that would preclude completion of the proposed study treatment at the opinion of the treating investigators.
3. Patients who are receiving any other investigational agents. Patients who have received other investigational agents previously who are no longer receiving these investigational agents may be eligible at the discretion of the PI.
4. Prior treatment with PD-1 inhibitors in the last 6 months or progression on a PD-1 inhibitor at any time.
5. Autoimmune disease or other pro-inflammatory conditions other than treated stable asthma, minor allergies (such as seasonal allergies), vitiligo or hypothyroidism.
6. Active and ongoing steroid use >10 mg prednisone, except for non-systemically absorbed treatments (such as inhaled or topical steroid therapy for asthma, COPD, allergic rhinitis).
7. Patients with uncontrolled intercurrent illness or any other significant condition(s) that would make participation in this protocol unreasonably hazardous, in the opinion of the Investigator.
8. Pregnant women are excluded from this study. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with breastfeeding should be discontinued if the mother is treated with pembrolizumab.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-12 (Estimated); Primary Completion 2030-12 (Estimated); Study Completion 2031-12 (Estimated)

PRIMARY OUTCOMES:
Dose Limiting Toxicity (DLT) Evaluation defined as the number of subjects experiencing a major, non-grade 5 adverse event as defined by CTCAE v6 or a grade 5 adverse event as defined by CTCAE 6. | From the initiation of study treatment to a minimum of 30 days following the end of active study treatment.
  To determine DLTs during Phase I to determine the recommended Phase 2 dose. A DLT is defined as experiencing ≥ Gr 4 AEs prior to surgery, a delay in surgery past 5 wks from RT, or ≥ Gr 4 surgical complications or Grade 5 adverse events are defined as deaths occurring during the study period, regardless of attribution, as assessed using CTCAE v6.0 criteria.
Major Pathologic Response (MPR) defined as less than 10% viable tumor on resected tumor specimen. | Surgery - Week 4
  To determine the major pathological response (MPR) in patients undergoing neoadjuvant X-ray photon radiation (XRT) or proton radiation (PT) with pembrolizumab followed by surgical salvage compared to a historical control group undergoing salvage surgery with PD-1 alone.

SECONDARY OUTCOMES:
Disease Free Survival as measured from time of surgery until either disease recurrence or death from any cause. | Surgery - Week 4 through 5 years
  To determine the disease-free survival (DFS) in patients undergoing neoadjuvant XRT or PT followed by surgical salvage compared to a historical control group undergoing salvage surgery alone. DFS is defined as the duration from time of surgery until either disease progression, recurrence or death due to any cause.
Safety using CTCAE v6.0 and toxicity evaluation. | 5 years
  To determine the safety of neoadjuvant pembrolizumab combined with XRT or PT prior to salvage surgery.

OTHER OUTCOMES:
Percent immune cell infiltration in tumors or microenvironment in patients undergoing neoadjuvant XRT or PT followed by surgical salvage determined by IHC and/or IF and/or Flow Cytometry. | Baseline (prior to radiotherapy) Cycle 1, Day 1 (Phase 1, post-radiotherapy) Cycle 1, Day 1 (Phase 2, post-radiotherapy and pembrolizumab initiation) Cycle 1, Day 22 Cycle 2, Day 1 Note: Neoadjuvant cycles are 28 days; adjuvant cycles are 42 days.
  To determine immunological changes in the tumor and microenvironment in patients undergoing neoadjuvant XRT or PT followed by surgical salvage.
Overall survival (OS) | 5 years
  To determine the overall survival (OS) in patients undergoing neoadjuvant XRT or PT and PD-1 followed by surgical salvage compared to a historical control group undergoing salvage surgery alone.
Overall response rate measured by RECIST criteria. | Week 4
  To determine the overall response rate by RECIST 1.1 after RT and PD-1.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Cincinnati Medical Center, Cincinnati, Ohio, United States

IPD SHARING:
Plan to Share IPD: Undecided